CLINICAL TRIAL: NCT03122665
Title: Effectiveness of Nefopam for Thermoregulation During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Laboratoires Biocodex (Montrouge, France) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 180/03
Record Dates: First submitted 2016-10-26; First posted 2017-04-21 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Hypothermia
Keywords: Nefopam; Pharmacokinetics; Shivering,; Thermoregulation; Anesthesia
MeSH Terms: conditions — Hypothermia | interventions — Nefopam

STUDY DESIGN:
Intervention Model Description: Volunteers given two doses of nefopam in a crossover protocol.
Who Masked: Participant, Investigator
Masking Description: Blinded drug containers.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nefopam low dose (Active Comparator): Nefopam continuous intravenous infusion at 0.5 mg/ml for three hours.
  Interventions: Drug: Nefopam Low dose
- Nefopam high dose (Active Comparator): Nefopam continuous intravenous infusion at 1.0 mg/ml for three hours.
  Interventions: Drug: Nefopam High dose

INTERVENTIONS:
Drug: Nefopam Low dose — Continuous intravenous infusion at 0.5 mg/ml for three hours.
  Other Names: Low
  Arms: Nefopam low dose
Drug: Nefopam High dose — Continuous intravenous infusion at 1.0 mg/ml for three hours.
  Other Names: High
  Arms: Nefopam high dose

SUMMARY:
Nefopam may help blunt thermoregulatory defenses, thus facilitating induction of therapeutic hypothermia

DETAILED DESCRIPTION:
Hypothermia, whether therapeutically induced or unintentional, triggers thermoregulatory defenses including vasoconstriction and shivering. Nefopam, a non-opioid, nonsteroidal centrally acting analgesic, has an opioid-sparing effect and anti-shivering potency without sedation, making it an ideal candidate to counteract thermoregulatory shivering.

Since complete compartmental pharmacokinetics (PK) are lacking this prospective, randomized, double-blind study in 8 volunteers was set to investigate the PK of arterial nefopam samples with non-linear mixed effect modelling. A two compartment mammillary model independent of covariates was found to describe the data best and could be implemented to drive automated pumps, achieving and maintaining a desired plasma concentration.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers ages 18-40

Exclusion Criteria:

* history of alcohol or drug abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
V1 | three hours of infusion
  Volume of distribution 1
V2 | three hours of infusion
  Volume of distribution2
CLel | three hours of infusion
  Clearance
CLdist | three hours of infusion
  Clearance distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, University of Bern, Bern, Freiburgstrasses, Switzerland

IPD SHARING:
Plan to Share IPD: No